CLINICAL TRIAL: NCT03537170
Title: Dietary Assessment and Prevalence of Refeeding Syndrome in High-risk TB Patients in Chhattisgarh, India
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201710162
Record Dates: First submitted 2018-05-11; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Tuberculosis; Refeeding Syndrome; Severe Malnutrition
MeSH Terms: conditions — Tuberculosis; Refeeding Syndrome; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe tuberculosis (TB) leads to wasting and anorexia, increasing risk of the refeeding syndrome (RFS) as defined by current criteria. TB patients have high metabolic rates and require a high calorie diet, with nutritional supplementation programs improving outcomes. BMI inversely correlates with mortality in these patients. Risk of RFS, a life-threatening syndrome associated with initiation of feeding after a period of low intake, has not been studied in this population and it is not known whether severely malnourished TB patients benefit from lower caloric intake. This study aimed to examine the prevalence of RFS in TB inpatients in rural India and correlate this with baseline and inpatient caloric intake.

ELIGIBILITY:
Inclusion Criteria:

* all adult inpatients admitted to the TB ward
* able to take enteral intake

Exclusion Criteria:

* unable to take enteral intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe tuberculosis patients admitted to the inpatient ward at Ganiyari hospital in Chhattisgarh, India.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Inpatient caloric intake | from date of admission to discharge, up to 100 weeks

SECONDARY OUTCOMES:
Incidence of refeeding syndrome | from date of admission to discharge, up to 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jan Swasthya Sahyog, Ganiyari, Chhattisgarh, India

IPD SHARING:
Plan to Share IPD: No